CLINICAL TRIAL: NCT02762799
Title: Single-center Open Randomized Clinical Trial to Evaluate Pharmacokinetics, Pharmacodynamics and Safety of Leucostim® (JSC "BIOCAD", Russia) Compared to Neupogen® (F. Hoffman-La Roche Ltd., Switzerland)
Brief Title: Clinical Trial to Evaluate Pharmacokinetics, Pharmacodynamics and Safety of Leucostim® Compared to Neupogen®
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Biocad (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: BCD-002-1
Record Dates: First submitted 2016-04-01; First posted 2016-05-05 (Estimated); Results first posted 2018-12-19 (Actual); Last update posted 2018-12-19 (Actual); Status verified 2018-12

CONDITIONS: Leucocytosis
Keywords: neutrophil count; filgrastim; granulocyte colony-stimulating factor
MeSH Terms: conditions — Leukocytosis | interventions — Filgrastim

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Leucostim® --> Neupogen®, subcutaneous injections (Experimental): Healthy volunteers in this group will receive single subcutaneous injection Leucostim® on Day 1 followed by single subcutaneous injection Leucostim® on Day 29.
  Interventions: Biological: Leucostim®; Biological: Neupogen®
- Neupogen® --> Leucostim®, subcutaneous injections (Experimental): Healthy volunteers in this group will receive single subcutaneous injection Neupogen®, on Day 1 followed by single subcutaneous injection Leucostim® on Day 29.
  Interventions: Biological: Leucostim®; Biological: Neupogen®
- Leucostim® --> Neupogen®, intravenous injections (Experimental): Healthy volunteers in this group will receive single intravenous injection Leucostim® on Day 1 followed by single intravenous injection Leucostim® on Day 29.
  Interventions: Biological: Leucostim®; Biological: Neupogen®
- Neupogen® --> Leucostim®, intravenous injections (Experimental): Healthy volunteers in this group will receive single intravenous injection Neupogen® on Day 1 followed by single subcutaneous intravenous Leucostim® on Day 29.
  Interventions: Biological: Leucostim®; Biological: Neupogen®

INTERVENTIONS:
Biological: Leucostim® — Leucostim® is filgrastim biosimilar.
  Other Names: filgrastim
Biological: Neupogen®
  Other Names: filgrastim

SUMMARY:
BCD-002-1 is 1 phase clinical trial to evaluate pharmacokinetics, pharmacodynamics and safety of single-injection of Leucostim® to healthy volunteers compared to Neupogen®

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent.
* Male gender.
* Age between 18 and 45 years.
* Normal body mass index.
* Verified diagnosis "healthy", established according to the anamnesis, physical examination and laboratory findings.
* Absence of alcohol or drug abuse.

Exclusion Criteria:

* History of use of filgrastim.
* Allergy to any components of study drugs.
* Acute hemorrhage, donation of blood / plasma or blood transfusions during last 2 months prior to enrollment in the study, history of chronic bleeding.
* Surgical interventions during last 30 days prior to screening or planed surgical intervention during the study.
* Any diseases that could interfere with pharmacokinetics of filgrastim, including chronic liver, liver or blood diseases, diseases of cardiovascular, lung and neuroendocrine systems.
* Fever with body temperature higher than 40°С.

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2016-07-18 (Actual); Primary Completion 2016-11-11 (Actual); Study Completion 2016-11-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Roman Ivanov, PhD, Study Chair — JCS BIOCAD

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Groups:
- Leucostim® --> Neupogen®, Subcutaneous Injections: Healthy volunteers in this group received single subcutaneous injection Leucostim® on Day 1 followed by single subcutaneous injection Leucostim® on Day 29.
  Leucostim®: Leucostim® is filgrastim biosimilar.
  Neupogen®
- Neupogen® --> Leucostim®, Subcutaneous Injections: Healthy volunteers in this group received single subcutaneous injection Neupogen®, on Day 1 followed by single subcutaneous injection Leucostim® on Day 29.
  Leucostim®: Leucostim® is filgrastim biosimilar.
  Neupogen®
- Leucostim® --> Neupogen®, Intravenous Injections: Healthy volunteers in this group received single intravenous injection Leucostim® on Day 1 followed by single intravenous injection Leucostim® on Day 29.
  Leucostim®: Leucostim® is filgrastim biosimilar.
  Neupogen®
- Neupogen® --> Leucostim®, Intravenous Injections: Healthy volunteers in this group received single intravenous injection Neupogen® on Day 1 followed by single subcutaneous intravenous Leucostim® on Day 29.
  Leucostim®: Leucostim® is filgrastim biosimilar.
  Neupogen®
Period: Overall Study
Arm/Group | Leucostim® --> Neupogen®, Subcutaneous Injections | Neupogen® --> Leucostim®, Subcutaneous Injections | Leucostim® --> Neupogen®, Intravenous Injections | Neupogen® --> Leucostim®, Intravenous Injections
Started | 18 | 18 | 12 | 12
Completed | 18 | 18 | 11 | 12
Not Completed | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Leucostim® --> Neupogen®, Subcutaneous Injections | Neupogen® --> Leucostim®, Subcutaneous Injections | Leucostim® --> Neupogen®, Intravenous Injections | Neupogen® --> Leucostim®, Intravenous Injections | Total
Number analyzed (Participants) | 18 | 18 | 12 | 12 | 60
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 22.94 [21.79 to 26.49] | 25.41 [22.45 to 29.58] | 23.48 [21.81 to 26.97] | 27.30 [24.61 to 27.78] | 24.63 [22.35 to 27.41]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0 | 0
  Male | 18 | 18 | 12 | 12 | 60
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: AUC (0-48 Hours)
Description: Area Under Curve (AUC) "concentration - time" from the moment of filgrastim injection to 48 hours
Time Frame: 0 to 48 hours post-dose
Measure: Geometric Mean (Standard Deviation); unit: picogram per ml / hour
Groups:
- Leucostim® Subcutaneous Injections: Healthy volunteers in this group received single subcutaneous injection Leucostim® on Day 1 (in Leucostim® --> Neupogen® group) or single subcutaneous injection Leucostim® on Day 29 (in Neupogen® --> Leucostim® group).
  Leucostim®: Leucostim® is filgrastim biosimilar.
  Neupogen®
- Neupogen® Subcutaneous Injections: Healthy volunteers in this group received single subcutaneous injection Neupogen®, on Day 1 (in Neupogen® --> Leucostim® group) or single subcutaneous injection Leucostim® on Day 29 (in Leucostim®-->Neupogen® group).
  Leucostim®: Leucostim® is filgrastim biosimilar.
  Neupogen®
- Leucostim® Intravenous Injections: Healthy volunteers in this group received single intravenous injection Leucostim® on Day 1 (in Leucostim® --> Neupogen® group) or single intravenous injection Leucostim® on Day 29 (in Neupogen®--> Leucostim® group)
  Leucostim®: Leucostim® is filgrastim biosimilar.
  Neupogen®
- Neupogen® Intravenous Injections: Healthy volunteers in this group received single intravenous injection Neupogen® on Day 1 (in Neupogen® --> Leucostim® group) or subcutaneous intravenous Leucostim® on Day 29 (in Leucostim®-->Neupogen® group)
  Leucostim®: Leucostim® is filgrastim biosimilar.
  Neupogen®
Arm/Group | Leucostim® Subcutaneous Injections | Neupogen® Subcutaneous Injections | Leucostim® Intravenous Injections | Neupogen® Intravenous Injections
Number analyzed (Participants) | 36 | 36 | 24 | 24
picogram per ml / hour | 168603.588 (47721.48) | 181152 (54706.439) | 411826.811 (204285.095) | 427355.99 (170878.6)

2. Primary Outcome: Cmax After Subcutaneous Injection
Description: Maximal concentration of filgrastim after subcutaneous injection of filgrastim
Time Frame: 0 to 48 hours post-dose
Measure: Geometric Mean (Standard Deviation); unit: picogram per ml
Arm/Group | Leucostim® Subcutaneous Injections | Neupogen® Subcutaneous Injections
Number analyzed (Participants) | 36 | 36
picogram per ml | 21605.163 (5247.467) | 23389.559 (7549.536)

3. Secondary Outcome: Cmax After Intravenous Injection
Description: Maximal concentration of filgrastim after intravenous injection of filgrastim
Time Frame: 0 to 48 hours post-dose
Measure: Geometric Mean (Standard Deviation); unit: picogram per ml
Arm/Group | Leucostim® Intravenous Injections | Neupogen® Intravenous Injections
Number analyzed (Participants) | 24 | 24
picogram per ml | 79751.577 (24810.907) | 90796.227 (25925.283)

4. Secondary Outcome: Tmax After Injection
Description: Time after single injection to reach maximal concentration of filgrastim
Time Frame: 0 to 48 hours post-dose
Measure: Median (Inter-Quartile Range); unit: hours
Arm/Group | Leucostim® Subcutaneous Injections | Neupogen® Subcutaneous Injections | Leucostim® Intravenous Injections | Neupogen® Intravenous Injections
Number analyzed (Participants) | 36 | 36 | 24 | 24
hours | 4 [4 to 4] | 4 [4 to 6] | 0.5 [0.5 to 2] | 0.5 [0.5 to 0.5]

5. Secondary Outcome: Т½
Description: Half-life of filgrastim after single injection of filgrastim
Time Frame: 0 to 48 hours post-dose
Measure: Median (Inter-Quartile Range); unit: hours
Arm/Group | Leucostim® Subcutaneous Injections | Neupogen® Subcutaneous Injections | Leucostim® Intravenous Injections | Neupogen® Intravenous Injections
Number analyzed (Participants) | 36 | 36 | 24 | 24
hours | 4,386 [3,889 to 4,914] | 4,307 [4,025 to 4,757] | 2,746 [2,178 to 2,951] | 2,549 [2,079 to 3,136]

6. Secondary Outcome: Kel
Description: The elimination rate constant after single injection of filgrastim
Time Frame: 0 to 48 hours post-dose
Measure: Mean (Inter-Quartile Range); unit: hour-1
Arm/Group | Leucostim® Subcutaneous Injections | Neupogen® Subcutaneous Injections | Leucostim® Intravenous Injections | Neupogen® Intravenous Injections
Number analyzed (Participants) | 36 | 36 | 24 | 24
hour-1 | 0.158 [0.141 to 0.173] | 0.161 [0.145 to 0.17] | 0.252 [0.173 to 0.318] | 0.272 [0.219 to 0.316]

7. Secondary Outcome: Clearance
Description: Clearance of filgrastim after single injection
Time Frame: 0 to 48 hours post-dose
Measure: Median (Inter-Quartile Range); unit: ml per hour
Arm/Group | Leucostim® Subcutaneous Injections | Neupogen® Subcutaneous Injections | Leucostim® Intravenous Injections | Neupogen® Intravenous Injections
Number analyzed (Participants) | 36 | 36 | 24 | 24
ml per hour | 2048.087 [1893.882 to 2518.863] | 1981.707 [1581.655 to 2439.947] | 965.938 [595.547 to 1055.471] | 830.442 [724.578 to 941.928]

8. Secondary Outcome: ANC-AUEC (0-336 Hours)
Description: Area Under Effect Curve (AUEC) "effect - time" from the moment of filgrastim injection to 336 hours based on absolute neutrophil count (ANC)
Time Frame: 0 to 336 hours post-dose
Measure: Geometric Mean (Standard Deviation); unit: cells х10^9 per liter/hour
Arm/Group | Leucostim® Subcutaneous Injections | Neupogen® Subcutaneous Injections | Leucostim® Intravenous Injections | Neupogen® Intravenous Injections
Number analyzed (Participants) | 36 | 36 | 24 | 24
cells х10^9 per liter/hour | 1924.284 (326.455) | 1933.358 (309.533) | 1860.922 (372.861) | 1895.82 (426.826)

9. Secondary Outcome: ANC-Emax
Description: Maximal absolute neutrophil count after single filgrastim injection
Time Frame: 0 to 336 hours post-dose
Measure: Geometric Mean (Standard Deviation); unit: cells х10^9 per liter
Arm/Group | Leucostim® Subcutaneous Injections | Neupogen® Subcutaneous Injections | Leucostim® Intravenous Injections | Neupogen® Intravenous Injections
Number analyzed (Participants) | 36 | 36 | 24 | 24
cells х10^9 per liter | 21.285 (4.593) | 20.803 (4.097) | 20.726 (6.393) | 21.602 (5.93)

10. Secondary Outcome: CD34-AUEC (0-336 Hours)
Description: Area Under Effect Curve (AUEC) "effect - time" from the moment of filgrastim injection to 336 hours based on CD-34 cells count (CD34)
Time Frame: 0 to 336 hours post-dose
Measure: Mean (Standard Deviation); unit: cell per microliter / hour
Arm/Group | Leucostim® Subcutaneous Injections | Neupogen® Subcutaneous Injections | Leucostim® Intravenous Injections | Neupogen® Intravenous Injections
Number analyzed (Participants) | 36 | 36 | 24 | 24
cell per microliter / hour | 1289 (762.292) | 1200.667 (761.29) | 1350.783 (716.645) | 1251.652 (562.087)

11. Secondary Outcome: CD34-Emax
Description: Maximal absolute count of CD34-cells after single filgrastim injection
Time Frame: 0 to 336 hours post-dose
Measure: Mean (Standard Deviation); unit: cell per microliter
Arm/Group | Leucostim® Subcutaneous Injections | Neupogen® Subcutaneous Injections | Leucostim® Intravenous Injections | Neupogen® Intravenous Injections
Number analyzed (Participants) | 36 | 36 | 24 | 24
cell per microliter | 7.694 (4.839) | 7.056 (5.248) | 9 (6.267) | 7.522 (4.22)

12. Secondary Outcome: Overall Frequency of Serious Adverse Events (SAE)
Time Frame: 0 to 336 hours post-dose
Measure: Count of Participants; unit: Participants
Arm/Group | Leucostim® Subcutaneous Injections | Neupogen® Subcutaneous Injections | Leucostim® Intravenous Injections | Neupogen® Intravenous Injections
Number analyzed (Participants) | 36 | 36 | 24 | 23
Participants | 0 | 0 | 0 | 0

13. Secondary Outcome: Overall Frequency of Adverse Events (AE)
Time Frame: 0 to 336 hours post-dose
Measure: Count of Participants; unit: Participants
Arm/Group | Leucostim® Subcutaneous Injections | Neupogen® Subcutaneous Injections | Leucostim® Intravenous Injections | Neupogen® Intravenous Injections
Number analyzed (Participants) | 36 | 36 | 24 | 23
Participants | 36 | 35 | 22 | 22

14. Secondary Outcome: Frequency of Local Reactions
Time Frame: 0 to 336 hours post-dose
Measure: Count of Participants; unit: Participants
Arm/Group | Leucostim® Subcutaneous Injections | Neupogen® Subcutaneous Injections | Leucostim® Intravenous Injections | Neupogen® Intravenous Injections
Number analyzed (Participants) | 36 | 36 | 24 | 23
Participants | 0 | 0 | 0 | 0

15. Secondary Outcome: Frequency of AE/SAE 3-4 Grade CTCAE 4.03
Description: Grading scale of CTCAE 4.03
  Grade refers to the severity of the AE. The CTCAE displays Grades 1 through 5 with unique clinical descriptions of severity for each AE:
  Grade 1 Mild; asymptomatic or mild symptoms; clinical or diagnostic observations only; intervention not indicated.
  Grade 2 Moderate; minimal, local or noninvasive intervention indicated; limiting age-appropriate instrumental ADL (activities of daily living).
  Grade 3 Severe or medically significant but not immediately life-threatening; hospitalization or prolongation of hospitalization indicated; disabling; limiting self care ADL.
  Grade 4 Life-threatening consequences; urgent intervention indicated. Grade 5 Death related to AE.
Time Frame: 0 to 336 hours post-dose
Measure: Count of Participants; unit: Participants
Arm/Group | Leucostim® Subcutaneous Injections | Neupogen® Subcutaneous Injections | Leucostim® Intravenous Injections | Neupogen® Intravenous Injections
Number analyzed (Participants) | 36 | 36 | 24 | 23
Participants | 0 | 1 | 0 | 0

16. Secondary Outcome: Frequency of Preliminary Withdrawal Due to AE/SAE
Time Frame: 0 to 336 hours post-dose
Measure: Count of Participants; unit: Participants
Arm/Group | Leucostim® Subcutaneous Injections | Neupogen® Subcutaneous Injections | Leucostim® Intravenous Injections | Neupogen® Intravenous Injections
Number analyzed (Participants) | 36 | 36 | 24 | 23
Participants | 0 | 0 | 0 | 0

17. Secondary Outcome: Proportion of Patients With Binding or Neutralizing Antibodies to Filgrastim
Description: Proportion of patients who had developed binding or neutralizing antibodies to filgrastim after single injection.
Time Frame: 0 to 336 hours post-dose
Measure: Count of Participants; unit: Participants
Arm/Group | Leucostim® Subcutaneous Injections | Neupogen® Subcutaneous Injections | Leucostim® Intravenous Injections | Neupogen® Intravenous Injections
Number analyzed (Participants) | 36 | 36 | 24 | 23
Participants | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Groups:
- Leucostim®, Subcutaneous Injections: Healthy volunteers in this group received single subcutaneous injection Leucostim® on Day 1(in group Leucostim®-->Neupogen®) or single subcutaneous injection Leucostim® on Day 29 (in group Neupogen® --> Leucostim®)
  Leucostim®: Leucostim® is filgrastim biosimilar.
  Neupogen®
- Neupogen® Subcutaneous Injections: Healthy volunteers in this group received single subcutaneous injection Neupogen®, on Day 1(in group Neupogen®-->Leucostim®) or single subcutaneous injection Neupogen® on Day 29 (in group Leucostim®-->Neupogen®)
  Leucostim®: Leucostim® is filgrastim biosimilar.
  Neupogen®
- Leucostim®, Intravenous Injections: Healthy volunteers in this group received single intravenous injection Leucostim® on Day 1(in group Leucostim®-->Neupogen®) or single subcutaneous injection Leucostim® on Day 29 (in group Neupogen® --> Leucostim®)
  Leucostim®: Leucostim® is filgrastim biosimilar.
  Neupogen®
- Neupogen®, Intravenous Injections: Healthy volunteers in this group received single intravenous injection Neupogen®, on Day 1(in group Neupogen®-->Leucostim®) or single subcutaneous injection Neupogen® on Day 29 (in group Leucostim®-->Neupogen®)
  Leucostim®: Leucostim® is filgrastim biosimilar.
  Neupogen®
Arm/Group | Leucostim®, Subcutaneous Injections | Neupogen® Subcutaneous Injections | Leucostim®, Intravenous Injections | Neupogen®, Intravenous Injections
All-Cause Mortality (participants affected / at risk) | 0/36 | 0/36 | 0/24 | 0/23
Serious Adverse Events (participants affected / at risk) | 0/36 | 0/36 | 0/24 | 0/23
Other Adverse Events (participants affected / at risk) | 36/36 | 35/36 | 22/24 | 22/23
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Leucostim®, Subcutaneous Injections (N=36) | Neupogen® Subcutaneous Injections (N=36) | Leucostim®, Intravenous Injections (N=24) | Neupogen®, Intravenous Injections (N=23)
Lymphocytosis (Blood and lymphatic system disorders) | 11 | 10 | 5 | 2
head pain (Nervous system disorders) | 9 | 10 | 0 | 0
Monocytosis (Blood and lymphatic system disorders) | 32 | 32 | 20 | 21
eosinophilia (Blood and lymphatic system disorders) | 10 | 15 | 9 | 7

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No